CLINICAL TRIAL: NCT04575571
Title: The MAVIPAN Protocol: For a Structured Response to the Psychosocial Consequences of the Restrictive Measures Imposed by the Global Health COVID-19 Pandemic
Brief Title: MAVIPAN: My Life and the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Collaborators: VITAM: Research Center on Sustainable Health (Unknown); Centre de recherche CERVO (Unknown); Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale (Other); Centre de recherche universitaire sur les jeunes et les familles (Unknown); Réseau québécois de recherche sur le vieillissement (Unknown); Participation sociale et villes inclusives (Unknown); Société inclusive (Unknown); CISSS de Chaudière-Appalaches (Other Government); Centre intégré de santé et de services sociaux de la Côte-Nord (Unknown); Fondation Mirella et Lino Saputo (Unknown); Ville de Québec (Unknown); Living Lab de Charlevoix (Unknown); Centre intégré de santé et de services sociaux du Bas St-Laurent (Unknown); Réseau provincial de recherche en adaptation réadaptation (Unknown); Réseau international sur le Processus de production du handicap (Unknown); Centre de recherche intégrée pour un système apprenant en santé et services sociaux (Unknown); Regroupement des organismes de personnes handicapées de la région 03 (Unknown)
Responsible Party: Principal Investigator, Annie Leblanc, Full Professor, Laval University
Other Study IDs: To be assigned
Record Dates: First submitted 2020-09-24; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Psychosocial Impacts of the COVID-19 Pandemic
Keywords: Psychological Distress; Coping Behaviors; Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention, this is an observational study that uses validated questionnaires and qualitative interviews.. — No intervention, this is an observational study that uses validated questionnaires and qualitative interviews.

SUMMARY:
The health crisis imposed by COVID-19 is forcing major worldwide social reorganization that will have profound consequences on our society. Currently, one-third of the world's population (~3 billion individuals) is living under some kind of isolation or quarantine measures, causing an unprecedented and rapidly evolving psychosocial crisis.

The psychosocial consequences of this health crisis will persist long after restriction measures are lifted and the pandemic is over. This impact will be significant for individuals facing unique contexts or challenges (e.g., older adults, individuals living with a disability, underprivileged families) and will most likely exacerbate existing social and gender inequalities in health and human development.

There is an urgent need for information on the evolution of the psychosocial dimensions of health and coping strategies used by our population and our health and social services structures. Thus, this study is designed to accelerate the availability of high-quality, real-time evidence within health and social services structures to address, support and minimize psychosocial consequences of the COVID-19 pandemic. Through constantly evolving research questions responsive to the course of the pandemic evolution, the rapid system transformations and adaptation of services, and knowledge users (KUs) needs, MAVIPAN aims to address, document, monitor, and evaluate the following:

1. Individuals and families' adjustments and mitigation strategies, especially for those considered vulnerable and in high-risk contexts.
2. Healthcare and social services workers and managers' adjustments and mitigation strategies.
3. The organization of service structures.
4. The social and economic response.

To achieve these objectives, we use a mixed methods study design that combines quantitative questionnaires and qualitative interviews to deepen our understanding of elements such as the coping strategies used during the pandemic. A first measure was taken during lock-down as well as a follow-up at 3 months. Another follow-up will be made at 7 months. At least one per year follow-up will be made over the course of the study (5 years). Additional measures may be taken depending on the evolution of the pandemic and the sanitary measures put in place by the authorities.

ELIGIBILITY:
Inclusion Criteria:

* General population

Exclusion Criteria:

* Not a resident of the province of Quebec
* Age under 14

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MAVIPAN is open to any individuals aged 14 and over across the Province of Quebec. We are particularly invested in recruiting vulnerable populations (e.g., older adults, individuals living with a disability or a chronic or mental health condition, child protection families, individuals living in institutional settings) and populations that have become vulnerable because of the COVID-19 context (e.g., healthcare and social services workers, adolescents, caregivers).
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2025-04-29 (Estimated); Study Completion 2025-04-29 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety and Stress Scale-21 (DASS-21) | Baseline (measured during lockdown in March 2020)
  The DASS-21 is a measure of depression, anxiety and stress symptoms. The score on each subscale varies from 0 to 21. A higher score means a higher level of symptoms.
Depression, Anxiety and Stress Scale-21 (DASS-21) | 3 months
  The DASS-21 is a measure of depression, anxiety and stress symptoms. The score on each subscale varies from 0 to 21. A higher score means a higher level of symptoms.
Depression, Anxiety and Stress Scale-21 (DASS-21) | 7 months
  The DASS-21 is a measure of depression, anxiety and stress symptoms. The score on each subscale varies from 0 to 21. A higher score means a higher level of symptoms.
Insomnia Severity Index | Baseline (measured during lockdown in March 2020)
  Scores vary between 0 and 28. A higher score means greater insomnia severity.
Insomnia Severity Index | 3 months
  Scores vary between 0 and 28. A higher score means greater insomnia severity.
Insomnia Severity Index | 7 months
  Scores vary between 0 and 28. A higher score means greater insomnia severity.
Warwick-Edinburgh Mental Well-Being Scale | Baseline (measured during lockdown in March 2020)
  Scores range from 7 to 35 and higher scores indicate higher positive well-being.
Warwick-Edinburgh Mental Well-Being Scale | 3 months
  Scores range from 7 to 35 and higher scores indicate higher positive well-being.
Warwick-Edinburgh Mental Well-Being Scale | 7 months
  Scores range from 7 to 35 and higher scores indicate higher positive well-being.
Hostility subscale- Symptoms Checklist-90-Revised | Baseline (measured during lockdown in March 2020)
  Only the Hostility subscale that measures thoughts, feelings and actions characteristic of anger is used. Scores range from 6 to 24 and higher scores indicate higher level of hostility
Hostility subscale- Symptoms Checklist-90-Revised | 3 months
  Only the Hostility subscale that measures thoughts, feelings and actions characteristic of anger is used. Scores range from 6 to 24 and higher scores indicate higher level of hostility
Hostility subscale- Symptoms Checklist-90-Revised | 7 months
  Only the Hostility subscale that measures thoughts, feelings and actions characteristic of anger is used. Scores range from 6 to 24 and higher scores indicate higher level of hostility
Substance use | Baseline (measured during lockdown in March 2020)
  These are self-report questions that measure the change in consumption level of different substances such as alcool, prescriptions medications and illicit drugs prior and after the lockdown.
Substance use | 3 months
  These are self-report questions that measure the change in consumption level of different substances such as alcool, prescriptions medications and illicit drugs prior and after the lockdown.
Substance use | 7 months
  These are self-report questions that measure the change in consumption level of different substances such as alcool, prescriptions medications and illicit drugs prior and after the lockdown.
Brief COPE | Baseline (measured during lockdown in March 2020)
  We use a subset of questions taken from the Brief Cope which measures coping strategies.
Dyadic Adjustment Scale | Baseline (measured during lockdown in March 2020)
  We use a subset of questions taken from the Dyadic Adjustment Scale which measures couple satisfaction.
Parental Stress Index | Baseline (measured during lockdown in March 2020)
  We only use the Interaction subscale which measures the extent to which the parent believes the child is not meeting expectations and finds interactions with the child are not reinforcing his parenting role.
Child Conflict Tactic Scale | Baseline (measured during lockdown in March 2020)
  We use a subset of questions that measures the presence of minor physical abuse as well as psychological abuse.
Strengths and Difficulties Questionnaire | Baseline (measured during lockdown in March 2020)
  We use a subset of questions that aim to measure different child behaviors and personality caracteristics.
Healthcare workers adaptation | Baseline (measured during lockdown in March 2020)
  We use a series of questions that assess different changes that may have occured in their work, as well as a series of beliefs they may hold concerning their work and their patients/clients.

CONTACTS AND LOCATIONS:
Overall Officials: Annie LeBlanc, PhD, Principal Investigator — Faculty of Medecine, Laval University
Locations (1):
- VITAM-Research Center in Sustainable Health, Québec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] LeBlanc A, Baron M, Blouin P, Tarabulsy G, Routhier F, Mercier C, Despres JP, Hebert M, De Koninck Y, Cellard C, Collin-Vezina D, Cote N, Dionne E, Fleet R, Gagne MH, Isabelle M, Lessard L, Menear M, Merette C, Ouellet MC, Roy MA, Saint-Jacques MC, Savard C; MAVIPAN Research Collaboration. For a structured response to the psychosocial consequences of the restrictive measures imposed by the global COVID-19 health pandemic: the MAVIPAN longitudinal prospective cohort study protocol. BMJ Open. 2022 Apr 4;12(4):e048749. doi: 10.1136/bmjopen-2021-048749. PMID 35379610
- See also: Official web site of the study — https://mavipan.ca/